CLINICAL TRIAL: NCT03790969
Title: Minimizing Pain Experience In Trigger Finger Steroid Injection.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, CHUAH SION KEAT, medical officer, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JEP-2018-654
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Trigger Finger
Keywords: steroid injection; pain; needle gauge; trigger finger
MeSH Terms: conditions — Trigger Finger Disorder; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 26 gauge needle (Experimental): intervention group
  Interventions: Device: 26 gauge needle
- 23 gauge needle (Active Comparator): control group
  Interventions: Device: 23 gauge needle

INTERVENTIONS:
Device: 26 gauge needle — smaller gauge needle
  Arms: 26 gauge needle
Device: 23 gauge needle — control group
  Arms: 23 gauge needle

SUMMARY:
To study the pain experience of trigger finger steroid injection with 26 gauge needle as compared to 23 gauge needle.

DETAILED DESCRIPTION:
compare pain experience of trigger finger steroid injection between 26 gauge needle and 23 gauge needle.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 year old
* Male or female(non-pregnant)
* Single trigger finger
* Clinically diagnosed trigger finger- Green classification Grade I or II
* No prior surgery to the involved finger
* Subject is able to provide voluntary, written informed consent

Exclusion Criteria:

* Age less than 18 year old
* Allergy to lignocaine or corticosteroid
* Trigger finger with Green classification grade III or IV
* Previous surgery on the affected finger
* Any wound, neurovascular injury, or skin disease at injection site
* Concomitant ipsilateral fingers/wrist/forearm/arm injury
* Preexisting congenital/acquired deformities of hand (such as rheumatoid arthritis, contracture)
* Insensate hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale-pain | one minute after injection
  A numerical rating scale of 0 to 100, with 0 meaning no pain and 100 meaning the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Chuah Sion Keat, Principal Investigator
Locations (1):
- Chuah Sion Keat, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No